CLINICAL TRIAL: NCT07127159
Title: Feasibility of a Music Listening Intervention for Mental Health Recovery in Chronic Stroke
Brief Title: Music Listening for Mental Health Recovery After Stroke
Acronym: IML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FY2024-8826
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: intentional music listening; music intervention; stroke; mental health; stroke recovery; music therapy; emotional well-being
MeSH Terms: conditions — Stroke; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intentional Music Listening (Experimental): Stroke patients assigned to the Intentional Music Listening group will participate in a 4-week intervention, in which participants will engage in one hour of music listening per day and complete daily self-reports on mood and control measures. Baseline, pre-, and post-intervention evaluations will assess clinical outcomes through behavioral measures of mental health and cognition. Pre- and post-intervention evaluations will also include biomarker assessments (MRI and physiological measures). The follow-up session will assess clinical outcomes only.
  Interventions: Behavioral: Intentional Music Listening
- Audiobook Listening (Active Comparator): Stroke patients assigned to the Audiobook Listening group will participate in a 4-week intervention, in which participants will engage in one hour of audiobook listening per day and complete daily self-reports on mood and control measures. Baseline, pre-, and post-intervention evaluations will assess clinical outcomes through behavioral measures of mental health and cognition. Pre- and post-intervention evaluations will also include biomarker assessments (MRI and physiological measures). The follow-up session will assess clinical outcomes only.
  Interventions: Behavioral: Audiobook Listening

INTERVENTIONS:
Behavioral: Intentional Music Listening — Participants will receive an iPad with Spotify (for music listening) and FaceTime. For 4 weeks (excluding weekends; 20 sessions), participants will listen to music for one hour per session, without multitasking (e.g., no chores or cooking), and will be encouraged to listen attentively. The investigators will collaborate with each participant to co-create a personalized playlist composed of self-selected, culturally relevant songs. This playlist can be updated at any time by the participant, either independently or with assistance from the team. During the music-listening session, participants will be on FaceTime with a team member, who will be available to provide support as needed. A custom Python script will continuously track the songs played by participants through Spotify, logging playback activity for research purposes.
  Arms: Intentional Music Listening
Behavioral: Audiobook Listening — Participants will be provided with an iPad equipped with a Spotify (for audiobook listening) and FaceTime. For 4 weeks (excluding weekends; 20 sessions), participants will be asked to listen to an audiobook of their choice for one hour per session, without engaging in other activities such as chores or cooking. Participants will be instructed to listen attentively and avoid multitasking during the session. A team member will connect with each participant via FaceTime to offer support. Participants may update or change their audiobook selections at any time, either independently or with help from the team. A custom Python script will be used to continuously track audiobook playback activity for research and analysis.
  Arms: Audiobook Listening

SUMMARY:
This study aims to explore whether listening to music intentionally can support the mental health of people recovering from a stroke. The question the investigators aim to answer is: Can intentional music listening improve emotional well-being in stroke survivors? And if so, what kinds of changes might music listening induce in mental health, thinking and memory (cognition), and brain activity? Participants will be randomly assigned to listen to either music or an audiobook for one hour each day, at home, for four weeks. Participants will also attend four in-person sessions with the researchers: at the start of the study (baseline), just before the listening period begins, after the four weeks are complete, and at a follow-up. During these visits, researchers will gather information about participants' mood and mental health (via questionnaires), assess memory and attention (via cognitive tasks), and use MRI scans to look at brain activity.

DETAILED DESCRIPTION:
This is a feasibility clinical trial of a remotely delivered music listening intervention for individuals with chronic stroke, incorporating objective tracking of music exposure and multimodal assessments of mental health, cognitive, neural, and physiological changes.

Specifically, this is a parallel-group randomized controlled feasibility trial enrolling patients with chronic stroke. Participants will be randomized to either an intentional music listening (IML) group or an active control group that listens to audiobooks. The study includes a 4-week pre-intervention period during which no treatment is administered; this phase is designed to assess the stability of outcome measures. Following this, participants will engage in 1-hour daily listening sessions over a 4-week intervention period. All listening activity (i.e., track identity, duration, and engagement) will be continuously tracked using custom open-source software, providing a measure of treatment dose. Behavioral outcomes related to mental health will be assessed at baseline, pre-intervention, post-intervention, and 3-month follow-up. Multimodal biomarkers (functional and structural MRI, electrodermal activity, and heart rate) will be collected pre- and post-intervention. The primary objective is to establish feasibility, defined by rates of retention and adherence, fidelity, feasibility, acceptability, and burden. Secondary outcomes include recruitment and randomization rates. This trial will provide essential data to inform the design of future large-scale clinical studies of IML for post-stroke mental health recovery.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 50 to 90
* Confirmed diagnosis of ischemic or hemorrhagic stroke occurring at least six months prior to enrollment.

Exclusion Criteria:

* Significant hearing loss, defined by a score >26 on the Hearing Handicap Inventory for the Elderly Screening (HHIE-S; Ventry and Weinstein, 1982)
* Contraindications for MRI
* Significant cognitive impairment, defined as a Montreal Cognitive Assessment (MoCA; Nasreddine et al., 2005) score below 22 (unless the lower score is attributable to expressive aphasia)
* Specific musical anhedonia, defined as a score below 60 on the Barcelona Music Reward Questionnaire (BMRQ; Mas-Herrero et al., 2013)
* Amusia, defined as a score below 70% on the Montreal Battery of Evaluation of Amusia (MBEA; Peretz et al., 2003).
* Participants will not be excluded if currently taking medications that may affect brain function (e.g., antidepressants) or if engaged in other complementary therapies (e.g., mindfulness, yoga). Participants will be allowed to initiate new medications or therapies during the study period.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Burden (Completion of evaluation sessions) | From baseline to follow-up (3 months post-intervention)
  Burden associated with each of the four evaluation sessions will be assessed. The outcome measure will include the proportion of patients who complete evaluations at each time point, with a target of at least 80% completion.
Burden Ratings | From baseline to follow-up (3 months post-intervention)
  Investigators will assess the perceived burden of participants by collecting at each evaluation session burden ratings. Participants will rate sessions as "not burdensome," "partially burdensome," or "very burdensome". The goal is for at least 80% of patients to rate the evaluations at each time point as "not burdensome. Burden ratings will be collected at 4 time points (baseline, pre-intervention, post-intervention and follow-up).
Patient acceptability | From beginning to end of the intervention (4 weeks)
  After each listening session, participants will rate the session as "not acceptable," "partially acceptable," or "fully acceptable." The goal is for at least 80% of sessions to be rated as fully acceptable.
Retention and Adherence | From beginning to end of the intervention (4 weeks)
  Proportion of enrolled and randomized participants who complete the IML/Audiobook sessions. At least 80% of randomized patients complete at least 80% of the IML/Audiobook sessions.
Feasibility Ratings | From beginning to the end of the intervention (4 weeks)
  Each listening session will be rated by the study team member leading the session as "not feasible," "partially feasible," or "fully feasible." The primary feasibility outcome measure is the proportion of sessions rated "fully feasible," with a target threshold of 80%.
Fidelity | From beginning to the end of the intervention (4 weeks)
  Fidelity will be measured as the the proportion of listening sessions delivered according to the protocol; video calls with patients will be recorded and a team member who was not present during the call will review the recordings and score the session as "delivered according to protocol" or "not delivered according to protocol". Benchmark for success: At least 80% of all sessions delivered according to the protocol.

SECONDARY OUTCOMES:
Recruitment | Baseline
  Recruitment will be measured by the number of participants successfully enrolled per month. The target benchmark is a minimum of 2 participants enrolled each month.
Randomization (Enrolment) | Baseline
  Randomization will be evaluated based on the proportion of screened participants who are successfully enrolled. The target benchmarks is for at least 30% of screened participants to be enrolled.
Randomization (Participation) | Baseline, pre-intervention, and intervention
  Randomization will be evaluated based on the proportion of enrolled participants who complete both the baseline and pre-intervention evaluations and attend at least one IML or Audiobook session. The target benchmark is for at least 80% of enrolled participants to reach this initial level of study engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ripolles, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Experimental data, devoid of any personal information, will be released as an open-source database.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol will be made available at the beginning of the trial (August 2025). All data will be available at the end of the trial (after fall 2026)
Access Criteria: Experimental data, devoid of any personal information, will be released as an open-source database. Access will be unrestricted.
URL: https://datadryad.org/

REFERENCES:
- [Background] Sihvonen AJ, Leo V, Ripolles P, Lehtovaara T, Ylonen A, Rajanaro P, Laitinen S, Forsblom A, Saunavaara J, Autti T, Laine M, Rodriguez-Fornells A, Tervaniemi M, Soinila S, Sarkamo T. Vocal music enhances memory and language recovery after stroke: pooled results from two RCTs. Ann Clin Transl Neurol. 2020 Nov;7(11):2272-2287. doi: 10.1002/acn3.51217. Epub 2020 Oct 6. PMID 33022148
- [Background] Baylan S, Haig C, MacDonald M, Stiles C, Easto J, Thomson M, Cullen B, Quinn TJ, Stott D, Mercer SW, Broomfield NM, Murray H, Evans JJ. Measuring the effects of listening for leisure on outcome after stroke (MELLO): A pilot randomized controlled trial of mindful music listening. Int J Stroke. 2020 Feb;15(2):149-158. doi: 10.1177/1747493019841250. Epub 2019 Apr 2. PMID 30940047
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Derived] Provias V, Kucukoglu MA, Robinson A, Yandun-Oyola S, He R, Palumbo A, Sihvonen AJ, Shi Y, Malgaroli M, Schambra H, Fuentes M, Ripolles P. Remote intentional music listening intervention to support mental health in individuals with chronic stroke: study protocol for a feasibility trial. BMJ Open. 2025 Sep 18;15(9):e109467. doi: 10.1136/bmjopen-2025-109467. PMID 40973376
- [Derived] Provias V, Kucukoglu MA, Robinson A, Yandun-Oyola S, He R, Palumbo A, Sihvonen AJ, Shi Y, Malgaroli M, Schambra H, Fuentes M, Ripolles P. Feasibility Trial Protocol for a Remote Intentional Music Listening Intervention to Support Mental Health in Individuals with Chronic Stroke. medRxiv [Preprint]. 2025 Aug 19:2025.08.15.25333806. doi: 10.1101/2025.08.15.25333806. PMID 40894150